CLINICAL TRIAL: NCT04727840
Title: Combined Dietary Intervention in Hyperkalemic CKD Patients With Potassium Binder (With Hyperkalemia) (DiPo Trial)
Brief Title: Potassium Binder in CKD Patients (With Hyperkalemia) (DiPo Trial)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lea Borgi, Associate Program Director, BWH/MGH Nephrology Fellowship Program Associate Physician, Renal Division, Brigham and Women's Hospital Instructor in Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000975
Record Dates: First submitted 2021-01-15; First posted 2021-01-27 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Diseases; Hyperkalemia
Keywords: Nutrition; Kidney Disease; Potassium binder; Sodium zirconium cyclosilicate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: Pilot study in 20 patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Other): All 20 CKD patients will be receiving a potassium binder while consuming a tailored diet of non-potassium restricted foods
  Interventions: Drug: Sodium Zirconium Cyclosilicate Oral Product

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate Oral Product — Sodium zirconium cyclosilicate (SZC), a non-absorbed cation exchanger, selectively binds potassium in the intestine. SZC is in a powder form and will be provided to patients in packets containing 5g or 10gm of the medication. Participants will mix the contents of one packet with water (about 45mL). The drink should be stirred and drank immediately. If powder remains in the glass, then water should be added and the remainder of the drink should be consumed. Other medications should be taken 2 hours before or after SZC.
  At Day 0 and Day 1, participants will be taking SZC at 10gm three times a day. A serum potassium will be checked on Day 2; if serum potassium is <5.1mEq/L, then the dose will be decreased to the maintenance dose of 5gm per day. At each serum potassium checks, the medication dosage will be adjusted accordingly.

SUMMARY:
This study hypothesizes that the administration of Sodium zirconium cyclosilicate in CKD patients with hyperkalemia while avoiding dietary potassium restriction will normalize their serum potassium levels. Additionally, we aim to assess the effects of a high potassium diet on renal function, endothelial function, acidosis, systemic inflammatory status and gut microbiota.

DETAILED DESCRIPTION:
A diet rich in fruits and vegetables is associated with better outcomes in CKD patients. However, the presence of hyperkalemia can prevent patients from increasing plant-based foods in their diets. While hyperkalemia can have severe health consequences in advanced CKD, the decreased consumption of plant-based foods can be associated with adverse health outcomes in this population.

Sodium zirconium cyclosilicate (SZC) is a non-absorbed cation exchanger that selectively binds potassium in the intestine.

This study plans to enroll CKD patients with an eGFR ≤45mL/min and a serum potassium ≥ 5mEq/L, administering SZC to achieve normokalemia, and provide them with a diet rich in fruits and vegetables. Endothelial function, inflammatory biomarkers and stool microbiota will be measured to assess the potential benefits of providing a diet rich in fruits and vegetables, albeit rich in potassium, in advanced CKD patients. Because these patients are usually restricting the intake of plant-based proteins and foods due to the concerns of hyperkalemia, eliminating this serious and potentially-life threatening clinical condition might carry health benefits, such as improved endothelial function and decreased inflammation

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18
* CKD stage 3-4 with an estimated GFR less or equal to 45 mL/min but greater than 15 mL/min
* Serum potassium level ≥5 mEq/L on two blood tests in the past 3 months but less than 6.5mEq/L

Exclusion Criteria:

* On dialysis
* Have been on SZC in the past 3 months
* Reside in a nursing home
* Pregnant patients
* Patients with known cognitive disability
* History of bowel disease such as but not limited to short bowel syndrome, bowel obstruction, inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
Normalization of Serum Potassium level | 2 days
  Achieve a serum potassium level less than 5mEq/L

SECONDARY OUTCOMES:
Change in Endothelial function | 15 days
  Improvement in endothelial function as measured by brachial artery ultrasound
Change in Acidosis (serum HCO3 levels) | 15 days
  Changes in acidosis measured by blood parameters
Systematic inflammatory status using serum biomarkers | 15 days
  Changes in inflammation measured by IL-6, CRP, Soluble urokinase-type Plasminogen Activator Receptor (suPAR), Monocyte Chemoattractant Protein-1 (MCP-1), Tumor Necrosis Factor Receptor (TNF-R), Fibroblast Growth Factor 23 (FGF23)
Changes in gut microbiota using stool collections | 15 days
  We will perform 16S rRNA sequencing from stool samples to determine microbiota diversity and species determination.

CONTACTS AND LOCATIONS:
Overall Officials: Lea Borgi, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No